CLINICAL TRIAL: NCT05560412
Title: Zein Nanoparticles for Glycemic Control
Acronym: GLUCOCAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022.152
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-11

CONDITIONS: PreDiabetes; Overweight and Obesity; Adult ALL
Keywords: Prediabetes; Glycemia and glucose metabolism; Zein; Glucose monitoring
MeSH Terms: conditions — Prediabetic State; Overweight; Obesity; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Randomised, double blind crossover intervention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The products (experimental and Placebo), will be produced by an external producer, who will retain the codes. None of the researchers involved in the study development or analyses will know the association until the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zein nanocapsules (Experimental): Subjects will consume daily a powder dissolved in water with nanoencapsulated zein
  Interventions: Dietary Supplement: Zein nanocapsules
- control (Placebo Comparator): Subjects will consume daily a powder dissolved in water with zein
  Interventions: Dietary Supplement: control

INTERVENTIONS:
Dietary Supplement: Zein nanocapsules — 1 g of Zein nanoencapsulated daily
  Arms: Zein nanocapsules
Dietary Supplement: control — 1 g of Zein non-encapsulated daily
  Arms: control

SUMMARY:
The use of zein nanoparticles as vehicles for drug delivery is under study, but of the effects observed in empty nanoparticles, in laboratory animals, the reduction of glucose levels was something worth studying. Thus, the present research on patients with prediabetes has been proposed. The objective is to assess the efficacy of zein nanoparticles on the glycemic control. For this purpose, a randomized, double blind crossover study has been designed.

Target sample size is 60.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obesity (BMI between 25 and 40 kg/m2
* Presence of prediabetes (fasting glycemia in blood between 100 and 126 mg/dL)
* No weight variations considered relevant (+/- 5%) in the last 3 months
* Metformin treatment is allowed, as far as dose is stable (at least 2 months with unvaried dose).
* Good physical and psychological state.

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Change in Fructosamine | 28 days
  Change in the levels of Fructosamine From day 0 to day 28
Change in GLP-1 AUC | Baseline, 15, 30, 45 and 60 minutes
  Change in AUC of postprandial GLP-1 levels after OGTT

SECONDARY OUTCOMES:
Fasting Plasma glucose | 28 days
  Change in Fasting Plasma glucose from day 0 to day 28
Continuous glucose levels | 28 days
  Area under the curve of 28 days of plasma glucose levels
Insulin Levels | 28 days
  Change in Fasting insulin levels from day 0 to day 28

OTHER OUTCOMES:
Cholesterol | 28 days
  Change in Total cholesterol from day 0 to day 28
HDL-Cholesterol | 28 days
  Change in HDL-cholesterol from day 0 to day 28
LDL-Cholesterol | 28 days
  Change in LDL-cholesterol from day 0 to day 28
Triglycerides | 28 days
  Change in Triglycerides from day 0 to day 28
Blood Pressure | 28 days
  Changes in DBP and SBP from beginning to end of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Investigacion en Nutricion. Universidad de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No